CLINICAL TRIAL: NCT05616299
Title: Human Clinical Trial to Evaluate the BRIGHTPOINT Reflectometer Device as Secondary Confirmation to Loss of Resistance in Lumbar Epidural Placement
Brief Title: BrightPoint Reflectometer Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Lumoptik, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY20220677
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Epidural Placement
Keywords: Labor; Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BrightPoint Epidural (Experimental): Subjects will receive an epidural using the BrightPoint device concurrent with usual LOR technique using the same epidural needle, sterile saline, syringe, etc.
  Interventions: Device: BrightPoint
- Normal Epidural (No Intervention): Subjects will have an epidural placed in usual manner with LOR technique using the same epidural needle, sterile saline, syringe etc. but without use of the BrightPoint device.

INTERVENTIONS:
Device: BrightPoint — Data from the BrightPoint device during epidural placement will be collected in real time on a tablet with pre-programmed software including tissue color and light reflectance with time stamps of when epidural space is entered as voiced by clinician per LOR.
  Arms: BrightPoint Epidural

SUMMARY:
Participants are being asked to participate in this study because they are having an epidural placed for labor. This human clinical trial has been designed to evaluate the use of the BrightPoint Reflectometer Device (AKA BrightPoint device) as secondary confirmation of Loss of Residence (LOR) for lumbar epidural placement by an experienced clinician. For this study, participants will be randomized to receive an epidural by an experienced clinician either with or without the use of the BrightPoint device. Epidurals performed as a part of this study will be done in a manner similar to how epidurals are currently performed in the hospital. The epidural space will be entered using usual loss of resistance technique for all patients. If the BrightPoint device is used, it will be as secondary verification of entry into the epidural space.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing an epidural procedure

Exclusion Criteria:

* Previous lumbar spine surgery
* Any known spinal abnormality that would interferre with successfully advancing a needle into the epidural space
* Any subject that requires an epidural needle longer than 4.0 inches
* Any procedure requiring use of CSE needles
* Any contraindication to neuraxial anesthesia
* No subjects in advanced active labor, e.g., 6-8 cm dilated
* Tattoo at the site of epidural insertion

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Number of times the BrightPoint device was able to measure Loss of Residence (LOR) accurately. | Up to 90 minutes
  This is measured as a Yes or No response.

SECONDARY OUTCOMES:
Number of times epidural accessed while using BrightPoint device as measured by clinical log | Up to 90 minutes
Number of times epidural catheter was used during the procedure as measured by clinical log | Up to 20 minutes
Number of adverse events as measured by clinician log | Up to 90 minutes
Number of times the BrightPoint device provided real-time secondary confirmation of Loss of Residence (LOR) as measured by clinician log | Up to 90 minutes
Number of times the BrightPoint device provided beneficial qualitative/quantitative clinical information to help complete the epidural as measured by clinician log. | Up to 90 minutes
Number of times clinician experienced the haptic feel of entering the ligamentum flavum (LF) as measured by clinician log | Up to 90 minutes
Number of times clinician experienced LOR after entering the epidural space as measured by clinician log | Up to 90 minutes
Number of times clinician experienced the haptic sensation of the needle contacting any tissue that was not expected as measured by clinician log | Up to 90 minutes
Number of times there were issues with catheterization as measured by clinician log | Up to 90 minutes
Number of times there were issues achieving pain management as measured by clinician log | Up to 4 hours
Number of times the device indicated the needle tip was entering the LF as measured by clinician log | Up to 20 minutes
Number of times the device showed a significant change of color from the light in LF to the dark in ES as measured by clinician log | Up to 90 minutes
Number of times the device showed a significant change of reflectance from high in LF to low in ES as measured by clinician log | Up to 90 minutes
Number of times the LOR and BrightPoint device agreed as measured by clinician log | Up to 90 minutes
Number of times coring was observed during procedure as measured by clinician log | Up to 90 minutes
Number of times the BrightPoint interfered with the ability to perform the epidural placement in the usual manner with LOR and haptic feedback as measured by clinician log | Up to 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lora Levin, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No